CLINICAL TRIAL: NCT03646292
Title: Comparison of The Effects of Thiazolidinediones(TZD), Sodium- Glucose Cotransporter 2 Inhibitors(SGLT2i) Alone and TZD / SGLT2i Combination Therapy on Metabolic Dysfunction-Associated Steatotic Liver Disease in Patients With Type 2 Diabetes
Brief Title: Antidiabetic Drugs for Steatotic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0655
Record Dates: First submitted 2018-08-10; First posted 2018-08-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Type 2 Diabetes; Digestive System Disease; Liver Diseases; Fatty Liver; Metabolic Dysfunction-Associated Steatotic Liver Disease; Non-Alcoholic Fatty Liver Disease; Hypoglycemic Agents; Physiological Effects of Drugs; Sodium-Glucose Cotransporter 2 Inhibitors; Pioglitazone; Molecular Mechanisms of Pharmacological Action; Empagliflozin; Thiazolidinediones
Keywords: Non-alcoholic Fatty Liver Disease; Hypoglycemic Agents; Physiological Effects of Drugs; Sodium-Glucose Cotransporter 2 Inhibitors; Pioglitazone; Molecular Mechanisms of Pharmacological Action; Empagliflozin; Metabolic Dysfunction-Associated Steatotic Liver Disease; Type 2 Diabetes; Digestive System Disease; Liver Diseases; Fatty Liver; Thiazolidinediones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Digestive System Diseases; Liver Diseases; Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone; empagliflozin

STUDY DESIGN:
Intervention Model Description: This study will evaluate the efficacy in lowering liver fat and the safety of empagliflozin 10mg, pioglitazone 15mg, alone or in combination (empagliflozin 10mg/pioglitazone 15mg), over a 24-week period.
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pioglitazone monotherapy (Experimental): Pioglitazone 15mg 1T daily for 24 weeks
  Interventions: Drug: Pioglitazone
- Empagliflozin monotherapy (Experimental): Empagliflozin 10mg 1T daily for 24 weeks
  Interventions: Drug: Empagliflozin
- Pioglitazone + Empagliflozin combination therapy (Experimental): Pioglitazone 15mg 1T + Empagliflozin 10mg 1T combination daily for 24 weeks
  Interventions: Drug: Combination of pioglitazone and empagliflozin

INTERVENTIONS:
Drug: Pioglitazone — The investigators will compare the degree of liver fat before and after pioglitazone monotherapy.
  Arms: Pioglitazone monotherapy
Drug: Empagliflozin — The investigators will compare the degree of liver fat before and after empagliflozin monotherapy.
  Arms: Empagliflozin monotherapy
Drug: Combination of pioglitazone and empagliflozin — The investigators will compare the degree of liver fat before and after pioglitazone and empagliflozin combination therapy.
  Arms: Pioglitazone + Empagliflozin combination therapy

SUMMARY:
To investigate the synergic therapeutic effect of thiazolidinediones and SGLT2 inhibitor on metabolic dysfunction-associated steatotic liver disease, the effect of empagliflozin 10mg, pioglitazone 15mg monotherapy and combination therapy in patients with type 2 diabetes and steatotic liver disease will be compared and analyzed.

This study was designed to include a total of 60 patients (20 per subgroup) for randomized controlled trials with prospective, open label, randomized, single-institution clinical trials.

The drug will be maintained for a total of 24 weeks. The primary endpoint is the difference of liver fat change measured by MRI-PDFF in the largest possible polygonal region of interest encompassing both lobes of the liver between three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 19 to 75 years
2. Individuals who are diagnosed with type 2 diabetes (HbA1c ≥ 7.5% and < 11.0%) and treated with antidiabetic drugs excluding TZD and SGLT2i over the previous 12 weeks
3. Individuals diagnosed with steatotic liver disease as documented by abdominal ultrasonography within the previous year
4. Individuals who have voluntarily agreed in written form to participate in the clinical trial after hearing the explanation of this clinical trial
5. Individuals who understand the content of the clinical trial and are able to participate in the trial until the end of the clinical trial

Exclusion Criteria:

1. Type 1 diabetes and gestational diabetes
2. Highly uncontrolled diabetes (HbA1c ≥ 11.0%)
3. Excessive alcohol intake (210 g and 140 g/week for men and women, respectively) within the previous 2 years
4. A history of taking thiazolidinedione or sodium-glucose cotransporter 2 inhibitor class medications within the last 12 weeks, or a history of discontinuing these medications due to severe side effects
5. Treatment with four or more classes of antidiabetic medications
6. Acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma, within 24 weeks
7. Intake of drugs that can cause steatotic liver disease (amiodarone, methotrexate, tamoxifen, valproate, etc.)
8. Allergy or hypersensitivity to the study drugs or their constituents
9. Oral or parenteral chronic corticosteroid therapy (more than 14 consecutive days) that requires continual adjustments in corticosteroid dose for therapeutic purposes within 8 weeks
10. Galactosemia
11. Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
12. Malignant tumors currently undergoing treatment or progression
13. A history of substance abuse or alcohol intoxication within 12 weeks
14. Infection of human immunodeficiency virus
15. Severe infection
16. Pre- and post-operative status, or severe trauma
17. Cardiac failure within 24 weeks (class III to IV in the NYHA classification)
18. Acute cardiovascular event within 12 weeks (unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass grafting, or coronary intervention)
19. AAcute and chronic renal disease (estimated glomerular filtration rate < 45 mL/min/1.73 m²) or dialysis
20. Pregnant or lactating women
21. Individuals whom the investigator determines to be unsuitable for participation in the clinical trial

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Change in liver fat fraction (%) measured by MRI-PDFF in the largest possible polygonal region of interest encompassing both lobes of the liver | After 24 weeks of treatment
  To measure the fat fraction, we drew the largest possible polygonal region of interest encompassing both lobes of the liver on a cross-sectional image, while avoiding blood vessels, bile ducts, and distinct hepatic lesions.

SECONDARY OUTCOMES:
Liver fibrosis measured by magnetic resonance elastography | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: liver stiffness (kPa) measured by magnetic resonance elastography.
The changes in lipid profile | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in lipid profile including total cholesterol (mg/dL), triglyceride (mg/dL), high-density lipoprotein-cholesterol (mg/dL), low-density lipoprotein-cholesterol (mg/dL), and free fatty acid (μEq/L).
The changes in liver enzyme | After 24 weeks of treatment
  he secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in liver enzyme including aspartate aminotransferase (IU/L), alanine aminotransferase (IU/L), alkaline phosphatase (IU/L), and gamma-glutamyl transferase (IU/L).
The changes in glucose metabolism | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in glucose metabolism including fasting glucose (mg/dL), HbA1c (%), fasting insulin (μIU/mL), homeostatic model assessment for insulin resistance (mg/dL*μIU/mL), and homeostasis model assessment of β-cell function (%)
The changes in cytokines | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in cytokines including high sensitivity C-reactive protein (mg/L), adiponectin (μg/mL), and leptin (ng/mL).
The changes in other biochemical parameters | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in other biochemical parameters including complete blood count, platelet count (10³/μL), total protein (g/dL), albumin (g/dL), total bilirubin (mg/dL), blood urea nitrogen (mg/dL), creatinine (mg/dL), and uric acid (mg/dL).
The changes in blood pressure and anthropometric parameters | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in blood pressure and anthropometric parameters including systolic and diastolic blood pressure (mmHg), body weight (kg), body mass index (kg/m², defined as weight [kg] divided by the square of the body height [m]), and waist circumference (cm).
The changes in body composition | After 24 weeks of treatment
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: The changes in body composition including abdominal subcutaneous fat area (cm²) and abdominal visceral fat area (cm²).
  To measure the body composition, abdominal fat content was assessed using a 3-mm thick cross-sectional abdominal fat CT scan at the midpoint of the L3 vertebra, with the participants in a supine position.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, 50-1 Yonsei-ro, Seodaemun-gu, Seoul 03722, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee M, Hong S, Cho Y, Rhee H, Yu MH, Bae J, Lee YH, Lee BW, Kang ES, Cha BS. Synergistic benefit of thiazolidinedione and sodium-glucose cotransporter 2 inhibitor for metabolic dysfunction-associated steatotic liver disease in type 2 diabetes: a 24-week, open-label, randomized controlled trial. BMC Med. 2025 May 7;23(1):266. doi: 10.1186/s12916-025-04017-x. PMID 40336058